CLINICAL TRIAL: NCT02105090
Title: Comparison of Novel Articaine Lozenge Versus Placebo for Upper Gastrointestinal Endoscopy in Adults. A Randomized Double-blinded Controlled Study
Brief Title: Efficacy Study of Articaine Lozenge to Enhance the Procedural Compliance of the Adults Undergoing Gastroduodenoscopy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Mihkel Meinberg, MD, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012-005528-13
Record Dates: First submitted 2014-03-29; First posted 2014-04-07 (Estimated); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Dyspepsia; Hematemesis; Abdominal Pain; Heartburn
Keywords: Upper gastrointestinal tract; Endoscopy; Lozenge; Articaine; Dyspepsia; Hematemesis; Abdominal pain; Heartburn
MeSH Terms: conditions — Dyspepsia; Hematemesis; Abdominal Pain; Heartburn | interventions — Anesthetics, Local; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sodium chloride 0.9% (Placebo Comparator): Sodium chloride 0.9% flavoured lozenge 10 ml administered orally (gargled and swallowed by patient) 3 minutes before the upper GI endoscopy
  Interventions: Drug: Sodium Chloride 0.9%
- Articaine hydrochloride 1% (Experimental): Articaine hydrochloride 1% flavoured lozenge 10 ml administered orally (gargled and swallowed by patient) 3 minutes before the upper GI endoscopy
  Interventions: Drug: Anesthetics, Local
- Articaine hydrochloride 2% (Experimental): Articaine hydrochloride 2% flavoured lozenge 10 ml administered orally (gargled and swallowed by patient) 3 minutes before the upper GI endoscopy
  Interventions: Drug: Anesthetics, Local

INTERVENTIONS:
Drug: Anesthetics, Local
  Other Names: Ultracain D ohne Adrenalin 20 mg/ml, ATC code N01BB08
  Arms: Articaine hydrochloride 1%; Articaine hydrochloride 2%
Drug: Sodium Chloride 0.9%
  Arms: Sodium chloride 0.9%

SUMMARY:
The purpose of this study is to examine in prospective, double-blinded randomised manner the ability of novel articaine-containing lozenge to enhance the procedure related compliance (compared to placebo) of the adult patients undergoing upper gastrointestinal endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* elective procedure
* weight over 40 kg
* American Society of Anesthesiology class I-III
* first upper GI endoscopy procedure
* finnish or/and swedish speaking

Exclusion Criteria:

* amide and/or esther local anaesthetic allergy
* paraben allergy
* Child-Pugh grade B/C liver failure
* renal insufficiency (calculated glomerular filtration rate under 60 ml/min/1.73 m2 according to Cockcroft-Gault scale )
* dementia
* those presenting with swallowing problem
* chronic pain condition
* chronic use of pain medication
* pregnancy
* lactation

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-10; Primary Completion 2019-12 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with 15% change in tolerability points according to Numeric Rating Scale (compared to baseline Numeric Rating Scale). | 30 minutes after the procedure

SECONDARY OUTCOMES:
Endoscopists´ procedural satisfaction points after the procedure assessed by using Numeric Rating Scale (NRS) | within 30 minutes after the procedure
Cumulative consumption of alfentanil during the procedure (mg) | 30 minutes after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Mihkel Meinberg, MD, Principal Investigator — Department of Anesthesiology and Intensive care medicine, Division of Surgery, Meilahti Hospital, Helsinki University Central Hospital; Reino Pöyhiä, MD, PhD, Study Chair — Department of Anesthesiology and Intensive care medicine, Division of Surgery, Meilahti Hospital, Helsinki University Central Hospital
Locations (1):
- Department of Anesthesiology and Intensive care medicine, Divison of Surgery, Meilahti hospital, Helsinki University Central Hospital, Helsinki, Uusimaa, Finland

REFERENCES:
- [Background] Campo R, Brullet E, Montserrat A, Calvet X, Moix J, Rue M, Roque M, Donoso L, Bordas JM. Identification of factors that influence tolerance of upper gastrointestinal endoscopy. Eur J Gastroenterol Hepatol. 1999 Feb;11(2):201-4. doi: 10.1097/00042737-199902000-00023. PMID 10102233
- [Background] Davis DE, Jones MP, Kubik CM. Topical pharyngeal anesthesia does not improve upper gastrointestinal endoscopy in conscious sedated patients. Am J Gastroenterol. 1999 Jul;94(7):1853-6. doi: 10.1111/j.1572-0241.1999.01217.x. PMID 10406247
- [Background] Shaoul R, Higaze H, Lavy A. Evaluation of topical pharyngeal anaesthesia by benzocaine lozenge for upper endoscopy. Aliment Pharmacol Ther. 2006 Aug 15;24(4):687-94. doi: 10.1111/j.1365-2036.2006.03023.x. PMID 16907901
- [Background] Evans LT, Saberi S, Kim HM, Elta GH, Schoenfeld P. Pharyngeal anesthesia during sedated EGDs: is "the spray" beneficial? A meta-analysis and systematic review. Gastrointest Endosc. 2006 May;63(6):761-6. doi: 10.1016/j.gie.2005.11.059. PMID 16650534
- [Background] Asante MA, Northfield TC. Variation in taste of topical lignocaine anaesthesia for gastroscopy. Aliment Pharmacol Ther. 1998 Jul;12(7):685-6. doi: 10.1046/j.1365-2036.1998.00355.x. PMID 9701534
- [Background] Mogensen S, Treldal C, Feldager E, Pulis S, Jacobsen J, Andersen O, Rasmussen M. New lidocaine lozenge as topical anesthesia compared to lidocaine viscous oral solution before upper gastrointestinal endoscopy. Local Reg Anesth. 2012;5:17-22. doi: 10.2147/LRA.S30715. Epub 2012 May 31. PMID 22915898
- [Background] Vree TB, Gielen MJ. Clinical pharmacology and the use of articaine for local and regional anaesthesia. Best Pract Res Clin Anaesthesiol. 2005 Jun;19(2):293-308. doi: 10.1016/j.bpa.2004.12.006. PMID 15966499
- [Background] Brinklov MM. Clinical effects of carticaine, a new local anesthetic. A survey and a double-blind investigation comparing carticaine with lidocaine in epidural analgesia. Acta Anaesthesiol Scand. 1977;21(1):5-16. doi: 10.1111/j.1399-6576.1977.tb01186.x. PMID 320810
- [Background] Kallio H, Snall EV, Luode T, Rosenberg PH. Hyperbaric articaine for day-case spinal anaesthesia. Br J Anaesth. 2006 Nov;97(5):704-9. doi: 10.1093/bja/ael222. Epub 2006 Aug 5. PMID 16891634
- [Background] Pitkanen MT, Xu M, Haasio J, Rosenberg PH. Comparison of 0.5% articaine and 0.5% prilocaine in intravenous regional anesthesia of the arm: a cross-over study in volunteers. Reg Anesth Pain Med. 1999 Mar-Apr;24(2):131-5. PMID 10204898
- [Background] Simon MA, Vree TB, Gielen MJ, Booij LH, Lagerwerf AJ. Similar motor block effects with different disposition kinetics between lidocaine and (+ or -) articaine in patients undergoing axillary brachial plexus block during day case surgery. Int J Clin Pharmacol Ther. 1999 Dec;37(12):598-607. PMID 10599952
- [Background] Vree TB, Baars AM, van Oss GE, Booij LH. High-performance liquid chromatography and preliminary pharmacokinetics of articaine and its 2-carboxy metabolite in human serum and urine. J Chromatogr. 1988 Feb 26;424(2):440-4. doi: 10.1016/s0378-4347(00)81126-3. No abstract available. PMID 3372637
- [Background] Prout BJ, Metreweli C. Pulmonary aspiration after fibre-endoscopy of the upper gastrointestinal tract. Br Med J. 1972 Nov 4;4(5835):269-71. doi: 10.1136/bmj.4.5835.269. PMID 4343464
- [Background] Oertel R, Rahn R, Kirch W. Clinical pharmacokinetics of articaine. Clin Pharmacokinet. 1997 Dec;33(6):417-25. doi: 10.2165/00003088-199733060-00002. PMID 9435991
- [Background] Simon MA, Vree TB, Gielen MJ, Booij LH. Comparison of the effects and disposition kinetics of articaine and lidocaine in 20 patients undergoing intravenous regional anaesthesia during day case surgery. Pharm World Sci. 1998 Apr;20(2):88-92. doi: 10.1023/a:1008622018161. PMID 9584343
- [Background] Alhashemi JA. Dexmedetomidine vs midazolam for monitored anaesthesia care during cataract surgery. Br J Anaesth. 2006 Jun;96(6):722-6. doi: 10.1093/bja/ael080. Epub 2006 Apr 4. PMID 16595611